CLINICAL TRIAL: NCT01984762
Title: Sleeve Gastrectomy and Roux-en-Y Gastric Bypass in the Treatment of Type 2 Diabetes Mellitus. Randomised Controlled Trial
Brief Title: Sleeve Gastrectomy and Roux-en-Y Gastric Bypass in the Treatment of Type 2 Diabetes Mellitus.
Acronym: CONTROL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 684-11
Record Dates: First submitted 2013-10-29; First posted 2013-11-15 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Type 2 Diabetes; Bariatric Surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RYGBP (Active Comparator): Roux-en-Y gastric bypass
  Interventions: Procedure: Roux-en-Y gastric bypass
- SG (Active Comparator): sleeve gastrectomy
  Interventions: Procedure: sleeve gastrectomy

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — RYGBP=Roux-en-Y gastric bypass
  Arms: RYGBP
Procedure: sleeve gastrectomy — SG = sleeve gastrectomy
  Arms: SG

SUMMARY:
Obesity is a growing epidemic throughout the world and is followed by increasing incidence of type 2 diabetes that accounts for 90-95% of all cases of diabetes. Weight loss is a major objective, although difficult to achieve with medical treatments. Many recent studies demonstrated that bariatric surgery has the potency to achieve marked and sustained weight loss, and is also associated with a significant improvement in control of type 2 diabetes. The principal aim of this study is to compare two types of bariatric procedures, the Roux-en-Y gastric bypass (RYGBP) and sleeve gastrectomy (SG). The study hypothesis is that these procedures have equal efficacy with regard to resolution of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus
2. BMI between 35 and 50kg/m2.
3. Males and females
4. Age between 18 and 60 years.

Exclusion Criteria:

1. Severe ongoing psychiatric disorder, alcoholism and substance abuse.
2. Redo operations after previous bariatric procedures.
3. Type 1 diabetes or other non-type 2 forms of diabetes
4. End stage renal disease, retinopathy, neuropathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Rate of resolution of type 2 diabetes | 5 years

SECONDARY OUTCOMES:
postoperative complications | 5 years
  Post-operative (within 30 days) bleeding, staple line/anastomotic leakage, infection, deep venous thrombosis, pulmonary embolism, resubmission. Questionnaires for health related quality of life (SF-36), gastroesophageal reflux symptoms (Carlsson-Dent), gastrointestinal symptom rating scale (GSRS) and food intake (SOS food questionnaire), recorded pre-operatively and at 6 weeks to 60 months post-operatively.

OTHER OUTCOMES:
Glycemic control mechanisms | 5 years
  Oral glucose tolerance tests comparing blood glucose, insulin and and other gastrointestinal hormone levels within and between the intervention groups pre- and post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fändriks, MD, PhD, Professor, Study Chair — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden